CLINICAL TRIAL: NCT05066490
Title: Effect of Exercise-induced Lipolysis on Vitamin D Status in Obese Children
Brief Title: Effect of Exercise on Vitamin d in Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Lamiaa Elsayyad, assistant professor, Taif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HAP-02-T-067 428
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Vitamin D Deficiency
MeSH Terms: conditions — Obesity; Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: 40 obese children who suffered from vitamin d deficiency were randomly assigned into three groups. group I (15 children) received endurance exercises and group II (15 children) received endurance exercises preceded by resistance exercises which have a stronger lipolytic effect. group III (10 children) acted as a control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endurance exercise (Experimental): This group received endurance exercises only.
  Interventions: Other: Endurance exercise
- resistance exersise plus endurance exersise (Experimental): This group received resistance exercises followed by endurance exercises.
  Interventions: Other: Endurance exercise; Other: Resistance exersises.

INTERVENTIONS:
Other: Endurance exercise — Treadmill training at moderate intensity.
Other: Resistance exersises. — Resistance exercises using the 10 repetition maximum.
  Arms: resistance exersise plus endurance exersise

SUMMARY:
The aim of the current study was to investigate the effect of exercise-induced lipolysis on vitamin D status in obese children. Two types of exercises that have different effects on lipolysis were used. Lipolysis was assessed via monitoring the level of plasma level of the free fatty acids and glycerol. Vitamin D was assessed through 25 (OH)D plasma levels.

DETAILED DESCRIPTION:
vitamin D status was monitored through 25 (OH)D levels, and the lipolysis status via the plasma level of the free fatty acids and glycerol immediately after the exercise. All subjects who participated in the study were under supervision for controlling the fat contents and vitamin D in their food for one week prior to the exercise. the subjects fasted eight hours before the exercise. All the exercises were performed between 9 am and 11 am.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index percentile equal to or greater than the 95th percentile
* All did not receive strength or balance training or involvement in competitive sports emphasizing muscular strength.
* All participants had balance deficiency and mobile flat foot.
* 25(OH) D was ranged from 10-20ng/ml

Exclusion Criteria:

* Injury to the lower limb required medical care.
* Deformity of or surgery in the lower limb.
* Visual impairment, or neuromuscular disorders.
* Engagement in obesity treatment programs, three months prior to the study.
* Epileptic fits
* Thyroid medications
* Autoimmune disease
* Take calcium or vitamin d3 supplements, medications for osteoporosis

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Free fatty acids | After 60 min of training
  Plasma level of the free fatty acids immediatlly after the exercise.
Glycerol | After 60 min of training
  Plasma level of glycerol immediatlly after the exercise.
Vitamin D | After 60 min of training
  Plasma level of 25 (OH) D immediatlly after the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem H Allam, Doctoral, Study Director — Assisstant professor
Locations (1):
- College of applied medical sciences, Ta'if, Mecca Region, Saudi Arabia